CLINICAL TRIAL: NCT01375725
Title: Mobius PT-INR Accuracy Clinical Study
Brief Title: Study to Determine the Accuracy of Prothrombin Time of Warfarinised Blood
Status: Completed | Type: Observational
Sponsor: Universal Biosensors Pty Ltd (Industry)
Responsible Party: Richard Ward, Assistant Professor, College of Pharmacy Harding University
Other Study IDs: MOB 0046
Record Dates: First submitted 2011-06-15; First posted 2011-06-17 (Estimated); Last update posted 2011-06-17 (Estimated); Status verified 2011-06

CONDITIONS: Clotting Disorders
MeSH Terms: conditions — Hemostatic Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Coumadin (warfarin): Subjects currently receiving coumadin (warfarin) treatment.

SUMMARY:
The purpose of this study is to measure prothrombin time (PT) expressed in International Normalised Ratio (INR) units in persons receiving coumadin (warfarin) treatment on an experimental device and a commercially available device. This study will involve taking a finger-puncture and testing onto a strip and meter system for the experimental and commercially available devices.

ELIGIBILITY:
Inclusion Criteria:

* Are currently taking coumadin (warfarin)
* Are aged 18 years or older
* Able and willing to provide informed consent
* Can understand (read and write) English
* Required to provide a capillary sample as part of their routine medical check

Exclusion Criteria:

* Previously participated in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects currently receiving coumadin (warfarin) treatment
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2010-09; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
PT/INR values from the experimental device will be statistically correlated to results obtained from a commercially available device | Five days to collect data and up to two weeks to generate correlation graph
  To determine the correlation of PT/INR values between an experimental and commercial device

CONTACTS AND LOCATIONS:
Overall Officials: Richard Ward, Pharm.D, Principal Investigator — Harding University
Locations (1):
- White River Diagnostic Clinic, Batesville, Arkansas, United States